CLINICAL TRIAL: NCT02121470
Title: The NGAL Test™ As An Aid for the Diagnosis of AKI in an Intensive Care Population, US
Brief Title: NGAL As An Aid for the Diagnosis of Acute Kidney Injury in Intensive Care
Status: Completed | Type: Observational
Sponsor: BioPorto Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: KLIN 12-005
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Acute Kidney Injury
Keywords: AKI; Acute Kidney Injury; Renal failure; NGAL; neutrophil gelatinase-associated lipocalin; lipocalin-2; siderocalin; Intensive care; ICU; Critical care
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, K3-EDTA Plasma, Li-Heparin Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute Kidney Injury (AKI) is a common and severe complication in critically ill patients which is associated with increased morbidity and mortality as well as high costs of medical care.

NGAL (neutrophil gelatinase-associated lipocalin, lipocalin-2, siderocalin) is a biomarker, that is expressed in several tissues including the kidneys. Renal expression of NGAL is dramatically increased in kidney injury from a variety of causes, and NGAL is released into both urine and plasma. NGAL levels rise within two hours of the insult, making NGAL an early and sensitive biomarker of kidney injury, with the potential to assist clinicians in managing patients at risk of kidney injury.

This study is designed to validate the assigned NGAL cutoff value by comparing to clinical diagnosis of AKI as determined by current clinical practice in the US.

The study sites will enroll consecutive ICU patients. Patients are given standard clinical care and lab-work. Each day, one additional urine and two additional plasma samples will be drawn and frozen. These additional samples are shipped to Sponsor for retrospective NGAL measurements.

The duration of each subject´s participation will be until discharge from the ICU, or for a maximum 8 days, whichever comes first. In addition serum creatinine values will continue to be collected manually from the hospital data system for 48 hours after discharge from the ICU. (If subject has been in ICU for 8 or more days, the follow up values are collected while the patient is still in the ICU).

250 subjects will be enrolled in total at the three investigator sites. At least 40 patients must be enrolled at each site.

The NGAL value will be matched to the "clinical diagnosis" of acute kidney injury (AKI) as specified by KDIGO® guidelines. The clinical diagnosis will be assigned by a three-person adjudication panel based on the entries in the eCRF by the investigators. Adjudicators are blinded for investigation site, AKI-diagnosis by treating physician, and NGAL values.

A comparison of AKI diagnosis based on the cutoff value 250 ng/mL and clinical diagnosis as assigned by the majority of the adjudication panel will be conducted.

DETAILED DESCRIPTION:
AKI is a common and severe complication in critically ill patients, which is associated with increased morbidity and mortality as well as high costs of medical care.

Despite efforts to standardize the definition and classification of AKI, there is still inconsistency in the application of the criteria and the limitations of serum creatinine and urine output for detecting AKI is generally recognized by the medical community. In the future, biomarkers of renal cell injury may identify additional patients with AKI and may identify the majority of patients at an earlier stage.

NGAL (neutrophil gelatinase-associated lipocalin, lipocalin-2, siderocalin) is such a biomarker. It is a small protein expressed in neutrophils and certain epithelia, including the renal tubules. Renal expression of NGAL is dramatically increased in kidney injury from a variety of causes, and NGAL is released into both urine and plasma. NGAL levels rise within two hours of the insult, making NGAL an early and sensitive biomarker of kidney injury.

Due to the heterogeneous implementation of AKI definitions and classifications, a uniform definition will be applied to this investigation, to ensure comparative results between the enrollment sites.

The aim of the study is to validate the assigned NGAL cutoff value by comparing to clinical diagnosis of AKI as determined by current clinical practice in the US.

The study sites will enroll consecutive patients meeting the criteria below in an ICU or critical care setting. Patients are given standard clinical care and lab-work. Each day, one additional urine and two additional plasma samples will be drawn and frozen. These additional samples are shipped to Sponsor for retrospective NGAL measurements.

The duration of each subject´s participation will be until discharge from the ICU, or for a maximum 8 days, whichever comes first. In addition serum creatinine values will continue to be collected manually from the hospital data system for 48 hours after discharge from the ICU. (If subject has been in ICU for 8 or more days, the follow up values are collected while the patient is still in the ICU).

250 subjects will be enrolled in total at the three investigator sites. At least 40 patients must be enrolled at each site.

The NGAL value will be matched to the "clinical diagnosis" of acute kidney injury (AKI) as specified by KDIGO® guidelines. The clinical diagnosis will be assigned by a three-person adjudication panel based on the entries in the eCRF by the investigators. Adjudicators are blinded for investigation site, AKI-diagnosis by treating physician, and NGAL values.

A comparison of AKI diagnosis based on the cutoff value 250 ng/mL and clinical diagnosis as assigned by the majority of the adjudication panel will be conducted.

.

Primary endpoints:

* Sensitivity of the NGAL test will be estimated as the proportion of patients with an observed NGAL value above or equal to 250 ng/ml among patients classified as having AKI, and.
* Specificity of the NGAL test will be estimated as the proportion of patients with an observed NGAL value below 250 ng/ml among patients classified as not having AKI

ELIGIBILITY:
Inclusion Criteria:

* Admission to intensive care unit
* Informed consent
* Age ≥ 18 years.

Exclusion criteria:

* History of nephrectomy, renal transplantation and/or renal replacement therapy initiated before admission
* Males and females aged 17 years or below

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care or critical care unit (all-comers)
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
NGAL (ng/mL) | Daily during ICU stay up to 8 days
  Highest measured value used

SECONDARY OUTCOMES:
Creatinine | Daily during ICU stay up to 8 days + 2 days after discharge
  Change from baseline/reference value calculated to be used in application of diagnostic AKI criteria and rating
Urine output | 6h, 12h and 24h daily during ICU stay up to 8 days
  Urine output calculated (mL/kg/h) to be used in application of diagnostic AKI criteria and rating

CONTACTS AND LOCATIONS:
Overall Officials: Peter A McCullough, M.D., Study Chair — St. John Providence Health System
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center / WNERTA, Springfield, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Methodist Hospital, Houston, Texas